CLINICAL TRIAL: NCT07104201
Title: An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Fenofibrate in Subjects With Primary Biliary Cholangitis (PBC)
Brief Title: Fenofibrate in Subjects With Primary Biliary Cholangitis (PBC)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252048-C-2
Record Dates: First submitted 2025-03-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fenofibrate (Experimental): Fenofibrate 200mg
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 200mg

SUMMARY:
An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Fenofibrate in Subjects with Primary Biliary Cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated)
2. Completed in a PBC study with fenofibrate(NCT06591455)
3. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

1. Treatment-related adverse event (AE) leading to study drug discontinuation in a previous PBC study with seladelpar
2. A medical condition, other than PBC, that in the Investigator's opinion would preclude full participation in the study or confound its results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Through study completion, up to 120 Months

SECONDARY OUTCOMES:
Normalization of ALP | 120 months
  Percentage of patients having normalization of ALP
Death | 120 months
  Occurrence of overall death
Liver transplantation | 120 months
  Occurrence of overall liver transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China